CLINICAL TRIAL: NCT07327216
Title: Efficacy and Safety of Sapylin Versus Dexamethasone Atomized Inhalation for Concurrent Chemoradiotherapy-Induced Oral Mucositis in Patients With Nasopharyngeal Carcinoma: A Randomized, Parallel, Non-inferiority Clinical Trial
Brief Title: Sapylin Versus Dexamethasone Inhalation for CCRT-Induced Oral Mucositis in Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PJKT2022-066
Record Dates: First submitted 2025-12-10; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Nasopharyngeal carcinoma; radiation-induced oral mucositis; Sapylin; Dexamethasone; atomized inhalation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — streptococcal preparation 722; Dexamethasone; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sapylin Group (Experimental): CCRT combined with Sapylin atomized inhalation (1 KE/time, QD from day 1 till the end of radiotherapy).
  Interventions: Drug: Sapylin; Combination Product: CCRT with Cisplatin
- Dexamethasone Group (Active Comparator): CCRT combined with Dexamethasone atomized inhalation (10 mg/time, QD from day 1 till the end of radiotherapy).
  Interventions: Drug: Dexamethasone; Combination Product: CCRT with Cisplatin

INTERVENTIONS:
Drug: Sapylin — Atomized inhalation, 1 KE/time, QD from day 1 of CCRT until the end of radiotherapy.
  Arms: Sapylin Group
Drug: Dexamethasone — Dexamethasone (10 mg per administration) via atomized inhalation once daily (QD).
  Arms: Dexamethasone Group
Combination Product: CCRT with Cisplatin — Patients receive cisplatin-based CCRT: cisplatin 80-100mg/m2, Q3W, three times during CCRT. Radiation dose: PTVnx: 69.96Gy/33F, PTV1: 60.06Gy/33F, PTV2: 54.12Gy/33F.

SUMMARY:
Radiation therapy is the main treatment for nasopharyngeal carcinoma (NPC), and standard care for advanced NPC often includes combination chemotherapy and radiation (CCRT). However, many patients experience serious side effects, such as painful mouth sores (Radiation-Induced Oral Mucositis, RTOM). These side effects can be so severe that they lower a patient's ability to adhere to treatment, potentially making the CCRT less effective. Studies have shown that a significant number of patients stop treatment early due to this toxicity.

Current clinical guidelines from organizations like MASCC/ISOO and ESMO agree that preventing RTOM is crucial, but there is currently no specific drug that works for everyone.

This study aims to investigate a new approach: using Sapylin, a biological immune regulator, delivered through an atomized inhaler. Preliminary research suggests Sapylin delivered this way may enhance the effectiveness of chemotherapy and boost the body's immunity.

The main purpose of this study is to determine the effect of Sapylin inhalation on the incidence and severity of RTOM, and to evaluate its safety and impact on the overall success of CCRT.

By participating, you will help researchers find a high-efficiency, low-toxicity method to improve CCRT outcomes and manage RTOM for future NPC patients and specialists.

ELIGIBILITY:
1. Inclusion Criteria:

   * Stage III-IVa NPC (AJCC 8th edition) diagnosed via pathology in a tertiary hospital;
   * No previous radiotherapy, chemotherapy, surgery, immunization, or targeted therapy;
   * Karnofsky Performance Status score ≥80;
   * Intact and normal oral mucosa before treatment;
   * Age 18-75 years;
   * Voluntary participation and provision of informed consent in person;
   * Routine blood examination: white blood cell count ≥4.0×109/L, hemoglobin ≥100g/L, neutrophil count ≥1.5×10^9/L, and platelet count ≥100×10^9/L;
   * Biochemical examination: total bilirubin ≤1.5×the upper limit of the normal range (ULN), alanine aminotransferase and aspartate aminotransferase ≤2×ULN, and estimated glomerular filtration rate ≥60 mL/min.
2. Exclusion Criteria:

   * With other malignant tumors in the past or present and/or distant metastasis during treatment;
   * Who have undergone surgery, chemoradiotherapy, and targeted immunotherapy;
   * With a history of asthma, rash, urticaria, and other allergic diseases;
   * With a history of autoimmune diseases, connective tissue diseases, and diabetes mellitus that significantly affect the healing of the oral mucosa;
   * With concomitant diseases, such as heart disease, kidney disease, and acute infectious diseases, which are judged by the investigator to seriously endanger the safety of patients or affect the completion of the study;
   * Who are breastfeeding, pregnant, or planning to become pregnant during the study;
   * With known allergies to the therapeutic agents and penicillin used in the trial;
   * Mental or nervous system diseases or poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Radiation-Induced Oral Mucositis (RIOM) | From the start of Concurrent Chemoradiotherapy (CCRT) through the completion of radiotherapy, assessed weekly for approximately 7 weeks.
  Incidence of RIOM is defined as the number of participants developing oral mucositis of any grade. Assessment is based on the World Health Organization (WHO) Oral Toxicity Scale. Scores range from 0 to 4 for ulceration, where higher scores indicate worse outcome.
Severity of Radiation-Induced Oral Mucositis (RIOM) | From Week 1 of Concurrent Chemoradiotherapy (CCRT) until the end of Radiotherapy (Week 7).
  To compare the severity of RlOM between the Sapylin and Dexamethasone groups using the World Health Organization (WHO) Oral Toxicity Scale. Scores range from 0 to 4 for ulceration, where higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Duration of Radiation-Induced Oral Mucositis (RIOM) | Daily assessment during CCRT, and up to 1 month after the completion of treatment (assessed up to 3 months).
  Time from the first diagnosis of RIOM (any grade) until the symptoms resolve to Grade 0 or return to baseline level.
Rate of Completion of Treatment Measures | Measured at the end of the concurrent chemoradiotherapy (CCRT) regimen (Week 7).
  Determined by comparing the actual dose and cycle count of Concurrent Chemoradiotherapy (CCRT) administered versus the planned total treatment regimen. Includes: 1) Actual dose divided by planned total dose (%); 2) Actual completed cycles divided by planned total cycles (%).
Incidence and Severity of Adverse Events (AEs) | Daily recording during treatment; Follow-up every 3 months for one year after treatment completion.
  All observed adverse events will be recorded and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Change in Body Mass Index (BMI) | Baseline (before CCRT starts) and at the end of treatment (End of Radiotherapy, approximately Week 7).
  Change is defined as the difference between BMI (kg/m2) at the end of treatment and baseline BMI (Baseline BMI: before CCRT starts).

CONTACTS AND LOCATIONS:
Overall Officials: Haiqing Luo, Principal Investigator — Specialty of Head and Neck Oncology, Affiliated Hospital of Guangdong Medical University
Locations (1):
- Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after study completion and publication.Data will be de-identified to protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after the study publication, extending for 3 years.
Access Criteria: Any investigator who submits a methodologically sound proposal will be granted access. The data will be de-identified individual participant data, and the purpose must be for scientific research.

REFERENCES:
- [Background] Peterson DE, Boers-Doets CB, Bensadoun RJ, Herrstedt J; ESMO Guidelines Committee. Management of oral and gastrointestinal mucosal injury: ESMO Clinical Practice Guidelines for diagnosis, treatment, and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v139-51. doi: 10.1093/annonc/mdv202. Epub 2015 Jul 4. No abstract available. PMID 26142468
- [Background] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Background] Kong D, Zhang D, Cui Q, Wang K, Tang J, Liu Z, Wu G. Sapylin (OK-432) alters inflammation and angiogenesis in vivo and vitro. Biomed Pharmacother. 2019 May;113:108706. doi: 10.1016/j.biopha.2019.108706. Epub 2019 Mar 4. PMID 30844656
- [Background] Nishii M, Soutome S, Kawakita A, Yutori H, Iwata E, Akashi M, Hasegawa T, Kojima Y, Funahara M, Umeda M, Komori T. Factors associated with severe oral mucositis and candidiasis in patients undergoing radiotherapy for oral and oropharyngeal carcinomas: a retrospective multicenter study of 326 patients. Support Care Cancer. 2020 Mar;28(3):1069-1075. doi: 10.1007/s00520-019-04885-z. Epub 2019 Jun 8. PMID 31177394

DOCUMENTS (2):
  • Study Protocol: Protocol Version V1.1 (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT07327216/Prot_002.pdf
  • Study Protocol and Informed Consent Form: Main Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT07327216/Prot_ICF_003.pdf